CLINICAL TRIAL: NCT01959685
Title: A Dose Escalating Study To Determine the Tolerability and Pharmacokinetics of a Single Dose of Androxal in Healthy Volunteers
Brief Title: A Dose Escalating Study to Determine the Tolerability and PK of a Single Dose of Androxal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA-109
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Pharmacokinetics; Tolerability
MeSH Terms: interventions — Enclomiphene; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalting (Experimental): Placebo, 125 mg Androxal, 250 mg Androxal each given as a single dose
  Interventions: Drug: Androxal; Drug: Placebo

INTERVENTIONS:
Drug: Androxal — 125 mg Androxal, 250 mg Androxal separated by at least 7 days
  Other Names: Enclomiphene citrate
Drug: Placebo — Placebo, single dose
  Other Names: Sugar pill

SUMMARY:
To determine the tolerability and pharmacokinetics (PK) of a single dose of Androxal in healthy adult male subjects as the dose to be investigated in a thorough QT interval/corrected QT interval (QT/QTc) study.

DETAILED DESCRIPTION:
A dose escalating study to determine the tolerability and pharmacokinetics (PK) of a supra-therapeutic dose of Androxal, up to 250 mg, in healthy adult male subjects as the dose to be investigated in a thorough QT interval/corrected QT interval (QT/QTc) study.

ELIGIBILITY:
Inclusion Criteria:

* Speaks, reads, and understands English or Spanish and is willing and able to provide written informed consent on an institutional review board (IRB)-approved form prior to the initiation of any study procedures;
* Male, between the ages of 18-60 years;
* No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
* Normal laboratory values (or abnormal but not clinically significant) at screening as determined by the Investigator;
* Subject is willing to remain in the clinic overnight for the Day 1 and Day 8 visits;
* Must be able to swallow gelatin capsules

Exclusion Criteria:

* Known hypersensitivity to Clomid;
* Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
* Subject with a significant organ abnormality or disease as determined by the Investigator;
* Any medical condition that would interfere with the study as determined by the Investigator;
* Slow cytochrome P450 2D6 (CYP2D6) metabolizer
* Participation in a clinical trial with investigational medication within 30 days prior to study medication administration;
* An acute illness within 5 days of study medication administration;
* Positive urine drug screen at the screening visit;
* A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
* History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
* History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of QTc interval prolongation;
* An employee or family member of an employee of the study site or the Sponsor;

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph S Podolski, Study Chair — Repros Therapeutics Inc.
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States

REFERENCES:
- See also: Sponsor corporate web site — http://www.reprosrx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Up to 250 mg Androxal: Subjects received a single dose each of placebo, 125 mg Androxal and 250 mg Androxal
Period: Overall Study
Arm/Group | Up to 250 mg Androxal
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Up to 250 mg Androxal
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics
Description: Cmax of a single dose 125 mg of Androxal
Time Frame: 24 hrs
Population: Safety population
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Up to 250 mg Androxal
Number analyzed (Participants) | 9
ng/dL | 11.0 (3.1)

2. Primary Outcome: Cmax of a Single Dose of 250 mg Androxal
Time Frame: 24 hours
Population: Safety population
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Up to 250 mg Androxal
Number analyzed (Participants) | 9
ng/dL | 24.9 (10.4)

ADVERSE EVENTS:
Time Frame: Up to 24 hours after last dose of study drug
Description: As all subjects received all treatments (placebo, 125 mg Androxal, and 250 mg Androxal, (adverse events could not be separated by treatment.
Arm/Group | Up to 250 mg Androxal
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Up to 250 mg Androxal (N=9)
Dermatitis contact (General disorders) | 1
Influenza like symptoms (Immune system disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights